CLINICAL TRIAL: NCT03482050
Title: A Phase I/IIa, Open Label, Dose-escalating Clinical Study to Evaluate the Safety, Tolerability and Theraputic Effects of Transplantation of Astrocytes Derived From Human Embryonic Stem Cells (hESC), in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate Transplantation of Astrocytes Derived From Human Embryonic Stem Cells, in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kadimastem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTRO-001-IL
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Dose-escalating, four subject-groups clinical study; a single treatment administration of AstroRx, administered in an escalating low, medium and high dose or two consecutive administrations of the medium dose separated by an interval. AstroRx will be administered by intrathecal (spinal) injection to subjects with ALS at the early disease stage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AstroRx (Experimental)
  Interventions: Biological: AstroRx

INTERVENTIONS:
Biological: AstroRx — Astrocytes derived from human embryonic stem cells

SUMMARY:
This is a study of transplantation of Astrocytes derived from human embryonic stem cells, in patients with Amyotrophic Lateral Sclerosis (ALS).

There will be no change in the routine ALS treatment of the patients enrolled into the study. Treatment will be administered in addition to the appropriate standard of care treatment.

The study hypothesis is that transplantation of Astrocyte(AstroRx) cells can compensate for the malfunctioning of patients' own astrocytes by restoring physiological capabilities like the reuptake of excessive glutamate, reducing oxidative stress, reducing other toxic compounds, as well as by secreting different neuroprotective factors

ELIGIBILITY:
Main Inclusion Criteria:

1. El Escorial criteria for probable or definite ALS
2. Males and and non pregnant females between 18 and 70 years of age
3. Patients with an ALS-FRS-R score of at least 30 with an ALS diagnosis of two years or less
4. No history of active psychiatric disorder. Patients receiving antidepressants as a preventive treatment, with no history of active psychiatric disorder may be included.
5. Patient has a good understanding of the study and nature of the procedure
6. Patient provides written informed consent prior to any study procedure
7. Patients should either be on a stable dose of Riluzole and/or Radicava® (if applicable) for at least 30 days, or not be treated with Riluzole and/or Radicava®
8. Patient is medically able to tolerate immunosuppression regimen
9. Presence of a willing and able caregiver who understands the need to attend all follow-up visits, even if mobility declines

Main Exclusion Criteria:

1. Patient has a past infection or a positive test for HBV,HCV or HIV
2. Patient is in need of respiratory support
3. Patient has a lower than 10/12 in ALS-FRS-R respiratory parameters or below 70% of predicted slow vital capacity (SVC)
4. Patient has renal failure
5. Patient has impaired hepatic function
6. Patient has a Body Mass Index (BMI) of <18.5 or > 30
7. Patient suffers from significant cardiac disease, diabetes, autoimmune diseases, chronic severe infection, malignant disease or any other disease or condition that may risk the patient or interfere with the ability to interpret the study results
8. Patient has systemic inflammation or active infections
9. Patient has been treated previously with any stem cell therapy
10. Current use of immunosuppressant medication or use of such medication within 6 weeks of Screening visit (Visit 0)
11. Patient has participated in another clinical treatment trial or received other experimental medications outside of a clinical trial within 1 month prior to start of this study
12. Any known immunodeficiency syndrome
13. Any concomitant disease or condition limiting patient safety to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by CTCAE Version 4.03 | 11 Months
  Safety and tolerability assessment will be based on treatment emerged adverse events

SECONDARY OUTCOMES:
Change in the ALS functional rating scale | 11 Months
  Preliminary efficacy assessment to measure response to treatment or progression of disease. Scale includes 12 questions related to tasks. Each task rated on a five-point scale from 0 = unable to do the task, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0 = worst and 48 = best.
Change in predicted slow vital capacity (%SVC) | 11 Months
  Preliminary efficacy assessment to measure respiratory muscle strength
Change in muscle strength grading by JAMAR grip strength | 11 Months
  Preliminary efficacy assessment to measure hand grip strength
Change in muscle strength grading by hand held dynamometer (HHD) | 11 Months
  Preliminary efficacy assessment to measure muscle strength in limb muscles
Change in Quality of Life questionnaire (ALSAQ-40) | 11 Months
  Preliminary efficacy assessment to measure the subjective well-being of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein Kerem Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Gotkine M, Caraco Y, Lerner Y, Blotnick S, Wanounou M, Slutsky SG, Chebath J, Kuperstein G, Estrin E, Ben-Hur T, Hasson A, Molakandov K, Sonnenfeld T, Stark Y, Revel A, Revel M, Izrael M. Safety and efficacy of first-in-man intrathecal injection of human astrocytes (AstroRx(R)) in ALS patients: phase I/IIa clinical trial results. J Transl Med. 2023 Feb 14;21(1):122. doi: 10.1186/s12967-023-03903-3. PMID 36788520